CLINICAL TRIAL: NCT07279493
Title: A Multicenter, Randomized, Double-Blind, Parallel, Placebo-Controlled Phase Ⅱb Clinical Trial to Evaluate the Efficacy and Safety of the KPCXM18 Injection at Different Doses in The Treatment of Acute Ischemic Stroke
Brief Title: Efficacy and Safety of the KPCXM18 Injection in Patients With Acute Ischemic Stroke
Acronym: KPCXM18
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kunming Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KPCXM18-C202; kyjtcrc (Registry Identifier: Duo Gao)
Record Dates: First submitted 2025-11-23; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low-dose group （The KPCXM18 injection） (Experimental): The KPCXM18 injection (60 mg BID)
  Interventions: Drug: The KPCXM18 injection
- high-dose group （The KPCXM18 injection） (Experimental): The KPCXM18 injection (100 mg BID)
  Interventions: Drug: The KPCXM18 injection
- Placebo (Placebo Comparator): Placebo of the KPCXM18 injection( BID )
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: The KPCXM18 injection — Intravenous infusion of 60 mg twice daily at intervals of 12±2 hours for 12±2 days.
  Arms: low-dose group （The KPCXM18 injection）
Drug: Placebo — Intravenous infusion twice a day with an interval of 12±2 hours for 12±2 days.
  Arms: Placebo
Drug: The KPCXM18 injection — Intravenous infusion of 100 mg twice daily at intervals of 12±2 hours for 12±2 days.
  Arms: high-dose group （The KPCXM18 injection）

SUMMARY:
This study is a multicenter, randomized, double-blind, parallel, placebo-controlled trial design to evaluate the efficacy and safety of the KPCXM18 injection at different doses for the treatment of acute ischemic stroke.

DETAILED DESCRIPTION:
Trial Objectives:

The primary objective is to evaluate the efficacy of the KPCXM18 injection at different doses for the treatment of acute ischemic stroke.

The secondary objective is to evaluate the safety of the KPCXM18 injection at different doses for the treatment of acute ischemic stroke and based on the population pharmacokinetic analysis method, explore the PK characteristics of the KPCXM18 injection in patients with acute ischemic stroke, and provide a basis for the design of the phase III clinical study.

Trial Design:

This trial is a multicenter, randomized, double-blind, parallel, placebo-controlled design. The subjects will be randomly assigned to the low-dose group, the high-dose group, and the placebo group at a ratio of 1:1:1, with 100 subjects in each group, totaling 300 subjects. The treatment will be administered continuously for 12±2 days to explore the efficacy and safety of the KPCXM18 injection at different doses for the treatment of acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18 to 80 years old (including 18 years old and 80 years old, based on the date of signing the informed consent form), male or female;
* 2.Diagnosed with acute ischemic stroke according to the " Chinese guidelines for diagnosis and treatment of acute ischemic stroke 2023 ";
* 3.During the screening process, it is required that the ischemic stroke should occur within 12 hours after the onset, and it is expected that the investigational drug can be started within 12 hours after the onset; note: The onset time is calculated from the time when the ischemic stroke symptoms appear, If the onset occurs during sleep, the time of onset should be considered as the last time the patient was observed to be normal;
* 4.Before intravenous thrombolysis, 6 points ≤ NIHSS score ≤ 24 points, and the sum of upper limb and lower limb score ≥2 points;
* 5.The patients who first attacked, or the patients who had a good prognosis after the last attacked , (mRS score was ≤1 before the onset of the disease );
* 6.The subject has received or plans to receive standard intravenous thrombolysis treatment after this onset;
* 7.The subject can understand and follow the research process and voluntarily signs the research informed consent form (the informed consent form is signed by the subject or the legal representative).

Exclusion Criteria:

* 1. Patients with intracranial hemorrhagic diseases confirmed by Imaging: hemorrhagic stroke, epidural hematoma, intracranial hematoma, subarachnoid hemorrhage, ventricular hemorrhage, Traumatic cerebral hemorrhage, etc;
* 2. Patients who have received or plan to receive endovascular interventional treatment (including endovascular mechanical thrombectomy, intravascular thrombus aspiration, arterial thrombolysis, angioplasty and stenting) or patients with arteriovenous bridging therapy after this onset;
* 3. Patients with disturbance of consciousness (NIHSS score Ia>1 point);
* 4. Patient has a history of intracranial hemorrhage before;
* 5. Patient who have a history of epilepsy or who experienced epileptic symptoms during a stroke;
* 6. The patient with other mental illness (such as severe mental disorders, dementia) and combined conditions such as limb movement disorders may influence their neurological function tests;
* 7. Patients with acute myocardial infarction, cardiac interventional therapy, or heart failure (grade III and IV according to NYHA) within the past 1 month;
* 8. Patients with malignant tumors, serious diseases of blood, digestion or other systems or diseases with bleeding tendencies (such as hemophilia, etc.), and the expected survival time is not more than 3 months;
* 9. Despite active antihypertensive therapy, hypertension remains uncontrolled: systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥100 mmHg;
* 10.Patients with severe liver function impairment, or ALT, AST > 2.0× ULN;
* 11.Patients with severe renal impairment, or serum creatinine > 1.5× ULN;
* 12.Patients who have used neuroprotective drugs (including Edaravone, Edaravone Dexborneol, Butylphthalide, Piracetam, Urinary Kallidinogenase, Ginkgolide, Ginkgo Diterpene Lactone, Safflower Extract and Aceglutamide Injection, etc.) after the onset of this illness;
* 13.Patients with severe allergies, hypersensitivity to at least two or more types of drugs, or known to be allergic to any ingredient or excipient of the investigational drug;
* 14.Patients with a history of major surgery within 1 month before screening;
* 15.Patients with a history of drug abuse within 3 month before screening;
* 16.Patients who participated in or are currently participating in other clinical trials within 3 month prior to this study;
* 17.Pregnancy, lactation. or patients who have a family plan within 3 months of the first dose and who are unwilling to use contraception;
* 18.The investigator considers that patients are not suitable for clinical trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-11-22 (Actual); Primary Completion 2026-10-18 (Estimated); Study Completion 2026-10-18 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS), with scores of 0-1 at Day 90 | day 90
  Proportion of subjects with mRS score ≤ 1 at day 90 after administration

SECONDARY OUTCOMES:
Modified Rankin Scale (mRS), with scores of 0-1 at day 12±2 and 30 | days 12±2 and 30
  Proportion of subjects with mRS score ≤ 1 at day 12±2 and 30 after administration
Modified Rankin Scale (mRS), with scores of 0-2 at days 12±2, 30 and 90 | days 12±2, 30 and 90
  Proportion of subjects with mRS score ≤ 2 at day 12±2, 30, 90 after administration
MRS Shift analysis | day 90
  MRS shift analysis at day 90 after administration
National Institute of Health stroke scale (NIHSS) on day 12±2 | days 12±2
  Proportion of subjects with NIHSS score ≤ 1 or with ≥4 point reduction from baseline at day 12±2 after administration
National Institute of Health stroke scale (NIHSS) on day 12±2 | days 12±2
  Change in NIHSS score from baseline at day 12±2 after administration
Barthel index (BI) at Day 90 | days 90
  Proportion of subjects with BI score ≥95 at day 90 after administration
Barthel index (BI) at Day 90 | days 90
  Proportion of subjects with BI score ≥75 at day 90 after administration

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (23):
- China (23):
  - Beijing Tiantan Hosptial，Capital Medical University, Beijing, Beijing Municipality
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Hengshui People's Hospital, Hengshui, Hebei
  - Da Qing Long Nan Hospital, Daqing, Heilongjiang
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - The People's Hospital Of Anyang City, Anyang, Henan
  - Nanshi Hospital Of Nanyang, Nanyang, Henan
  - Nanyang Second General Hospital, Nanyang, Henan
  - The First Affiliated Hospital Of Nanyang Medical College, Nanyang, Henan
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Meihakou Central Hospital, Meihekou, Jilin
  - Affiliated Central Hospital Of Shenyang Medical College, Shenyang, Liaoning
  - The First People's Hospital Of Shenyang, Shenyang, Liaoning
  - The People's Hospital Of Liaoning Province, Shenyang, Liaoning
  - Yan'an University Xianyang Hospital, Xianyang, Shaanxi
  - First People's Hospital Of Tancheng, Linyi, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - Tengzhou Central People's Hospital, Tengzhou, Shandong
  - Sinopharm Tongmei General Hospital, Datong, Shanxi
  - Linfen Central Hospital, Linfen, Shanxi
  - Linfen People's Hospital, Linfen, Shanxi
  - Jiaxing Second Hospital, Jiaxing, Zhejiang

IPD SHARING:
Plan to Share IPD: No